CLINICAL TRIAL: NCT05996887
Title: Impact of Enhanced Recovery After Surgery (ERAS) for Sleeve Gastrectomy on Postoperative Nausea and Vomiting: Controlled Randomized Study.
Brief Title: Impact of ERAS on Postoperative Nausea and Vomiting After Sleeve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, haidy salah mansour, assistant professor of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 820:6/2023
Record Dates: First submitted 2023-07-29; First posted 2023-08-18 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Nausea and Vomiting, Postoperative
Keywords: sleeve gastrectomy; nausea; vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non- enhanced recovery after surgery (Placebo Comparator): All patients will receive antiemetics as haloperidol 2 mg and dexamethasone 8 mg and ondansetron 8 mg in addition to standard care protocol.
  Interventions: Other: standard care protcol
- enhanced recovery after surgery (Active Comparator): All patients will receive antiemetics as haloperidol 2 mg and dexamethasone 8 mg, and ondansetron 8 mg in addition to following the recommendation of ERAS society guidelines.
  Interventions: Other: enhanced recovery protocol

INTERVENTIONS:
Other: standard care protcol — All patients will receive antiemetics as haloperidol 2 mg and dexamethasone 8 mg and ondansetron 8 mg in addition to standard care protocol.
  Other Names: control
  Arms: non- enhanced recovery after surgery
Other: enhanced recovery protocol — All patients will receive antiemetics as haloperidol 2 mg and dexamethasone 8 mg and ondansetron 8 mg in addition to following the recommendation of ERAS society guidelines.
  Other Names: ERAC
  Arms: enhanced recovery after surgery

SUMMARY:
The use of bariatric surgery in the treatment of severe obesity has several benefits in terms of sustainable weight loss, improvements, or resolution of several metabolic comorbidities as well as improved life expectancy.

Gastric surgery, history of acid reflux and reduction in gastric size, in particular after laparoscopic sleeve gastrectomy (LSG), surgery may further contribute to postoperative nausea and vomiting (PONV).

The combination of antiemetic drugs that act at different receptors is more effective than using only one drug in preventing PONV in patients with increased risk for these events.

DETAILED DESCRIPTION:
After obtaining Institutional Ethical Committee approval and written informed consent from the patients in each case, the ASA score, Simplified Apfel scores14 a measure of PONV risk, and duration of preoperative fasting are calculated for each patient. Patients will be randomly allocated into two groups.

Group 1 (non-ERAS): All patients will receive haloperidol 2 mg, dexamethasone 8 mg, and ondansetron 8 mg in addition to standard care protocol.

Group 2 (ERAS): All patients will receive haloperidol 2 mg, dexamethasone 8 mg, and ondansetron 8 mg in addition to following the recommendation of ERAS society guidelines.

All patients will receive general anesthesia. The doses of anesthetic drugs for induction and maintenance of anesthesia are calculated with reference to the ideal body weight (IBW) and the corrected body weight (CBW) in patients, where IBW=height (in cm)-100 for men and height (in cm)-105 for women and CBW=IBW+ [0.4 × (current weight-ideal weight)]12.

Anesthesia and Operative Technique for Non-ERAS:

1. Anesthesia:

   Induction of anesthesia IS carried out with propofol 2 mg kg -1 iv of CBW, fentanyl 3 μg kg-1 CBW, and cisatracurium 0.1 mg kg-1 iv of IBW for tracheal intubation. The maintenance IS performed with fentanyl 0.1 to 0.3 μg kg-1 min -1 iv of IBW, isoflurane 1 % mixture of oxygen and air 1:1, and an additional dose of cisatracurium if necessary. Neuromuscular blockade IS reversed with neostigmine up to 0.04 mg kg-1 IV of IBW and atropine up to 0.015 mg kg-1 iv of IBW.
2. Antiemetic protocol:

   * Dexamethasone 8mg IS administered 90 min prior to induction of anesthesia.
   * Haloperidol 2 mg after induction of anesthesia and ondansetron 8 mg IS infused 20 to 30 min prior to the end of the operation.
3. Postoperative Analgesia Analgesia IS done with intravenous ketorolac 30 mg immediately after the induction of anesthesia and maintained at 8 h and acetaminophen IV 1 g every 6 h. IS used in the PACU to keep PVRS<4. Patient-controlled analgesia (PCA) containing 20 mg Nalbuphine (Nalbuphine HCl 20mg / 1ml) to 100 ml with normal saline over 24 hours. The PCA infuser unit IS infused at a rate of 2 ml.h-1 with a lockout time of 15 min & bolus of 1 ml per time. The intensity of pain IS measured by a pain verbal rating scale (PVRS, 0=no pain to 10=worst pain)12.

Anesthesia and Operative Technique for ERAS:

The institutional ERAS is described in Table 1. Table 1: Technique for ERAS15,16. Preoperative protocols

Pain management • Acetaminophen 1000mg PO 2h before anesthesia

* Gabapentin 400 ml PO before anesthesia Diet • Clear liquids until 3 h prior to surgery PONV prevention • H2 receptor antagonist
* Dexamethasone 8mg IS administered 90 min prior to induction of anesthesia Preoperative fasting
* Fasting to solids until 6 h before induction and clear liquids until 2 h before induction.

Intraoperative protocols

Anesthesia General anesthesia: TIVA16,17

* Propofol (2 mg kg-1 iv of CBW). GA IS maintained with i.v. infusion of propofol (75-150 mg kg-1 min-1).
* Dexmedetomidine (0.5 mg kg-1 i.v. over 10 min) IS initiated and maintained with an i.v. infusion of dexmedetomidine (0.1-0.3 mg kg-1h-1).
* Ketamine a single dose before incision (0.5 mg kg-1 i.v.) then 0.5 mg.kg-1.h-1.
* Muscle relaxation with cisatracurium 0.1 mg kg-1 iv of IBW IS maintained with boluses additional dose of cisatracurium if necessary. Neuromuscular blockade IS reversed with neostigmine up to 0.04 mg kg-1 IV of IBW and atropine up to 0.015 mg kg-1 iv of IBW.
* Patients are ventilated with a mixture of oxygen and air. At the end of the surgery, muscle relaxation IS reversed with neostigmine (up to 5 mg) and glycopyrrolate (0.2-0.8 mg).

Antiemetic protocol: • Haloperidol 2mg IS administered immediately after induction of anesthesia and ondansetron IS infused 20 to 30 min prior to the end of the operation.

Pain management • Lidocaine 1 mg kg, then by 1 mg kg-1 hr-1. continuous infusion 1 mg. kg -1h-1. for maintenance.

* Magnesium Sulfate (30 mg/kg) + continuous infusion (10 mg/kg/h)
* Bilateral Transversus Abdominis plane block (TAP) at the end of the operation. Fluid management • Goal-directed IV fluid therapy, avoiding both restrictive or liberal strategies.

Abdominal drainage and nasogastric decompression • Nasogastric tubes and abdominal drains should not be used Postoperative protocols Pain management • Bilateral Transversus Abdominis plane block (TAP) at the end of the operation.

* Lidocaine IV drip for 24 h
* Acetaminophen IV transitioned to PO.
* Ketoralac 30 mg every 8 h
* acetaminophen IV 1 g every 6 h.
* IV Nalbuphine, breakthrough pain. The intensity of pain IS measured by a pain verbal rating scale (PVRS, 0=no pain to 10=worst pain)

PONV treatment • Ondansetron 8 mg IS used as the primary rescue antiemetic and metoclopramide 10 mg IV IS utilized in PONV refractory to ondansetron.

Thromboprophylaxis

* Thromboprophylaxis should involve mechanical and pharmacological measures. Doses and duration of treatment should be individualized.

Fluid management • Stop IV fluids on POD 1 Early postoperative nutritional care • Stop IV fluids on POD 1

• Clear liquids on POD 0 PO: Per oral, PONV: postoperative nausea and vomiting, IV: intravenous, prn: when required, POD: postoperative day.

Postoperative Care for both groups:

1. Feeding A liquid diet IS prescribed for the first postoperative day, followed by a diet containing broth without residue as tolerated by the patient.
2. Rescue Antiemetic The PONV IS defined as at least one episode of nau¬sea, vomiting, or retching. PONV IS evaluated as follows: I = no nausea or vomiting, II = nausea but no vomiting, III = mild to moderate vomiting, and IV = severe and frequent vomiting more than five times within 24h.

   The severity of postoperative nausea (PON) IS assessed using a numeric rating scale (I = mild, II = mod¬erate, III = severe).

   The severity of postoperative vomiting (POV) IS recorded according to the number of vomiting episodes (I = no vomiting, II = vomiting episodes occurring 1-2 times within 24 h, III = vomiting episodes occurring 3-5 times within 24 h, IV = vomiting episodes occurring more than 5 times within 24 h). The volume of postoperative water intake IS measured during the two periods (0-24 h and 24-36h). Nausea IS assessed hourly during the first two hours, every two hours for the following four hours, and every four hours until the 24th hour. Nausea IS evaluated on a three-point scale from 0 (no nausea), 1 (mild nausea) to 2 (severe nausea). A patient IS classified to have had PONV if any nausea and/or vomiting occurred within the first 24 postoperative hours.

   The patient IS given ondansetron IV as the primary rescue antiemetic and metoclopramide 10 mg IV IS utilized in PONV refractory to ondansetron, when there IS an episode of vomiting or if there IS a request at any time made by the patient for treatment of symptoms.
3. Outcome Variables Secondary endpoints included time to first administration of rescue antiemetic drug, the number of rescues, postoperative opioid consumption, time to tolerate oral fluid, and time to readiness for discharge. Data collection IS done by blinded personnel at the end of the following postoperative time intervals: 0-2, 2-12, 12-24, and 24-36 h, postoperatively. The quality of recovery IS assessed by QoR-1518 questionnaires at discharge. In patients who are discharged before 36 h, the questionnaires are filled out during a telephone call the next morning.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years

* Sex: Both sex
* ASA Physical Status: II, III.
* Body mass index: Between 40 and 60 kg/m2.
* Participants: Patients who are undergoing elective Sleeve Gastrectomy

Exclusion Criteria:

* Patients with hypersensitivity or contraindication to haloperidol, dexamethasone, or ondansetron.
* Serious complications in the perioperative period (such as shock, cardiac arrest, hemorrhage, needing transfusion).
* Psychiatric disorder.
* History of migraine.
* Use of opioid, hormonal, anti-inflammatory, and antiemetic medication 24 h prior to surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-30 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative nausea and vomiting | 36 hours
  number and percentage of episode of nausea and vomiting
  : I = no nausea or vomiting, II = nausea but no vomiting, III = mild to moderate vomiting, and IV = severe and frequent vomiting more than five times within 24h.
  The severity of postoperative nausea (PON) was assessed using a numeric rating scale (I = mild, II = mod¬erate, III = severe).

SECONDARY OUTCOMES:
Time to first administration of rescue antiemetic drug. | 36 hours
  Time in minute
postoperative opioid consumption. | 36 hours
  amount in ml of opioid given in the 36 hours after surgery
Time to tolerate oral fluid | 36 hours
  time in minute
The quality of recovery. | 36 hours
  questionnaire: QoR 15 patient survey
complications. | 36 hours
  number and percentage of complication related to technique of TAP as hematoma formation at the injection site, vascular or lymphatic injury, neurologic symptoms and local anesthetic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: haidy S mansour, MD, Principal Investigator — Assistant professor
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No